CLINICAL TRIAL: NCT02065414
Title: Four Weeks Clinical Efficacy of an Ethyl Lauroyl Arginate HCL (LAE) Mouth Rinse: Effect on Gingivitis
Brief Title: A Clinical Trial to Test the Effect of Experimental Mouth Rinse on Gum Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: LAEBBA0005
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Gingivitis
Keywords: Gums; Gingiva; Gingival Inflammation; Gingival Bleeding
MeSH Terms: conditions — Gingivitis; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neg Control Mouth Rinse W002194-0221-P (Placebo Comparator): Mouth rinse containing 5% Hydroalcohol
  Twice each day, brush in usual manner with a fluoride-containing dentifrice, rinse mouth with water, and then rinse with 20 ml of mouth rinse W002194-0221-P for 30 seconds and spit it out.
  Interventions: Other: Mouth rinse containing 5% Hydroalcohol
- Experimental: Mouth Rinse 19668-012 (Experimental): Listerine Advance Gum Defense Twice each day, brush in usual manner with a fluoride-containing dentifrice, rinse mouth with water, and then rinse with 20 ml of mouth rinse 19668-012 for 30 seconds and spit it out - do not swallow.
  Interventions: Other: Listerine Advance Gum Defense
- Active Comparator Mouth Rinse 5000347078873 (Active Comparator): Mouth rinse containing Chlorhexidine Corsodyl ®Mouthwash
  Twice each day, brush in usual manner with a fluoride-containing dentifrice, in the usual manner, rinse mouth with water, wait 5 minutes after brushing and then rinse with 10 ml of mouth rinse 5000347078873for 60 seconds and spit it out - do not swallow.
  Interventions: Other: Mouth rinse containing Chlorhexidine

INTERVENTIONS:
Other: Listerine Advance Gum Defense
  Arms: Experimental: Mouth Rinse 19668-012
Other: Mouth rinse containing Chlorhexidine
  Arms: Active Comparator Mouth Rinse 5000347078873
Other: Mouth rinse containing 5% Hydroalcohol
  Arms: Neg Control Mouth Rinse W002194-0221-P

SUMMARY:
Participants will be given special instructions about taking care of their teeth during the 18 hours before they come to the dentist's office for screening/baseline, 1 week, 2 weeks and 4 weeks. At that first visit, they will be examined by a dentist, who will examine their mouths with a dental instrument to determine whether they qualify to participate in the trial. Someone who works for the dentist will also take some oral measurements.

Participants who qualify to be in the study will receive a treatment for their gingivitis and have an equal chance of being assigned to one of three treatment groups. Participants in all three groups will be given toothpaste that is already available in stores. They will brush their teeth twice daily in their regular manner. After brushing, participants in one group will use an experimental mouth rinse that is not available in stores. Another group will be given a mouth rinse to use that is already available in stores, and the third group will use a placebo mouth rinse. After they receive their assigned products participants will be supervised while they brush their teeth and rinse to ensure they understand exactly how to use the products. Participants will be required to stay at the site 20 minutes after the first use of product during visit 1 to monitor any potential allergic reaction. All other brushing and rinsing over the next four weeks will be at home, but participants will be required to keep a diary to record their brushing and rinsing times twice each day.

Participants will be required to bring their diaries and any left-over toothpaste and mouth rinse with them for three more scheduled appointments after about 1 week, 2 weeks, and 4 weeks. At those appointments, the dentist will examine their mouths, make sure there are no safety concerns, and examine again to get the measurements needed. One of the dentist's staff members will take other measurements as well.

The study will determine the measured effects of the experimental mouth rinse on bleeding as a result of gingivitis, and compare these results to the mouth rinse that is already available.

DETAILED DESCRIPTION:
At screening Participants will present to the clinical site having refrained from oral hygiene for at least 8 hours, but no more than 18 hours for baseline examinations (safety oral and hard soft tissue exam, MGI - Modified Gingival Index, BI - Bleeding Index and PI- Plaque Index and Extrinsic Staining. After the baseline oral examinations, qualifying participants will receive a whole-mouth supragingival dental prophylaxis and will be randomly assigned to one of three treatment groups.

Participants randomly assigned to the negative control treatment group will brush twice daily with a marketed fluoride toothpaste in their usual manner and rinse with a placebo mouth rinse. Participants randomly assigned to the experimental treatment group will brush twice daily with a marketed fluoride toothpaste brush in their usual manner and use an experimental mouth rinse. The last treatment group randomly assigned to the positive control will brush twice daily with a marketed fluoride toothpaste in their usual manner and rinse with a marketed available mouth rinse. Participants will have an equal chance of being assigned each of the three groups. The first product use will be conducted under supervision of study personnel. Participants will be required to stay at the site 20 minutes after the first use of product during visit 1 to monitor any potential analytic reaction. All other brushing and rinsing will be unsupervised and the participants will be required to maintain a diary card to document twice-daily product use, brushing and rinsing times. Diaries along with product accountability will be used to check for subject compliance.

Participants will return to the clinical site after 1 week (Day 7±1 day), 2 weeks (Day 14±2 days) and 4 weeks (Day 28±3 days). Oral hard and soft tissue safety, Modified Gingival Index (MGI), Bleeding Index (BI), and Plaque Index (PI) will be assessed by the primary examiner 1 at all visits Extrinsic stain will be assessed at baseline, 2 weeks and 4 weeks by the secondary examiner.

At the end of the study, subjects will return all used and unused product to the clinical site.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females 18 years of age or older, in good general and oral health without any known allergy to commercial dental products or cosmetics.
* 2. Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial and all questions have been answered.
* 3. Females of childbearing potential must be using a medically-acceptable method of birth control for at least 1 month prior to Visit 1 and agree to continue using this method during their participation in the study.
* 4. Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel's assessment.
* 5. A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count.
* 6. A mean gingival index ≥1.75 according to the Modified Gingival Index.
* 7. A mean plaque index ≥1.95 according to the Turesky modification of the Quigley-Hein Plaque Index scored on six surfaces per tooth.
* 8. Mean Bleeding Index ≥0.15
* 9. Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator.
* 10. Absence of moderate/advanced periodontitis based on a clinical examination (ADA Type III, IV).
* 11. Absence of fixed or removable orthodontic appliance or removable partial dentures.

Exclusion Criteria:

* 1. History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes and mouth rinses and red food dye.
* 2. Dental prophylaxis within 2 weeks prior to Screening visit.
* 3. History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
* 4. Antibiotic, anti-inflammatory or anticoagulant therapy during the study or within the one month prior to the baseline exam. Intermittent use of certain anti-inflammatory medication is acceptable at the discretion of the investigator.
* 5. Daily use of aspirin.
* 6. Known sensitivity to the investigational product ingredients.
* 7. Self reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).
* 8. Significant unstable or uncontrolled medical condition which may interfere with a subject's participation in the study, at the discretion of the Investigator.
* 9. Participation in any clinical study within 30 days of Visit 1.
* 10. Relative, partner or staff of any clinical research site personnel.
* 11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Whole Mouth Mean Bleeding Index (BI) at 4 weeks | 4 weeks
  Bleeding will be assessed by using a standard measurement called the Gingival Bleeding Index.

SECONDARY OUTCOMES:
Whole Mouth Mean Bleeding Index (BI) at 1 week | Within 2 weeks
  Bleeding will be assessed by using a standard measurement called the Gingival Bleeding Index
Whole-mouth Mean Modified Gingival Index (MGI) | Within 4 weeks
  Gingivitis will be assessed by scoring inflammation according to the Modified Gingival Index.
Turesky Modification of the Quigley Hein Plaque Index (PI) | Within 4 weeks
  Plaque will be assessed using a standard scale called the Turesky Modification of the Quigley Hein Plaque Index
Extrinsic Stain | Within 4 weeks
  Stain will be assessed using the standard measurement called Macpherson Modification of the Lobene Stain Index

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, DMD, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- National Research Ethics Committee Yorkshire & Humber-Sheffield, Chester, United Kingdom, United Kingdom